CLINICAL TRIAL: NCT01589510
Title: A Study of Lumigan® 0.01% in Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/034
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumigan® 0.01%: Lumigan® 0.01% (bimatoprost 0.01% ophthalmic solution) as prescribed by physician per standard practice for up to 14 weeks.
  Interventions: Drug: bimatoprost 0.01% ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost 0.01% ophthalmic solution — Bimatoprost 0.01% ophthalmic solution (Lumigan® 0.01%) as prescribed by physician per standard practice for up to 14 weeks.
  Other Names: Lumigan® 0.01%

SUMMARY:
A study of Lumigan® 0.01% as administered in standard practice for patients with POAG or OHT. All treatment decisions, care and diagnostic procedures provided are at the discretion of the participating physicians according to their clinical judgment and the local standard of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG or OHT
* Prescribed Lumigan® 0.01%

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with POAG and OHT
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumigan® 0.01%
Started | 419
Completed | 386
Not Completed | 33

BASELINE CHARACTERISTICS:
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 419
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18 to 30 years | 1
  31 to 40 years | 7
  41 to 50 years | 33
  51 to 60 years | 66
  61 to 70 years | 137
  71 to 80 years | 116
  81 to 90 years | 51
  >=91 years | 4
  Missing | 4
Sex/Gender, Customized [Number; unit: Participants]
  Female | 232
  Male | 183
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Baseline
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eyes at Baseline.
Time Frame: Baseline
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 390
Millimeters of Mercury (mmHg)
  Right Eye | 21.23 (4.72)
  Left Eye (n=389) | 21.38 (4.51)

2. Secondary Outcome: Physician Evaluation of IOP Lowering in the Study Eye(s)
Description: IOP is a measurement of the fluid pressure inside the eye. Physicians evaluated IOP compared to the target IOP for each patient's study eye(s). The numbers of eyes in each category are presented.
Time Frame: Week 14
Population: All patients with data for this outcome measure
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 391
Number analyzed (Eyes) | 436
Eyes
  IOP lower than target | 83
  Target IOP reached | 233
  IOP decreased but target not reached | 73
  IOP increased | 6
  No change | 13
  Data Missing | 28

3. Secondary Outcome: Patient Assessment of Tolerability on a 4-Point Scale
Description: Patient assessment of tolerability was assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: Week 14
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 393
Patients
  Very Good | 201
  Good | 167
  Moderate | 16
  Poor | 9

4. Secondary Outcome: Physician Assessment of Tolerability on a 4-Point Scale
Description: Physician assessment of tolerability was assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: Week 14
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 392
Patients
  Very Good | 209
  Good | 171
  Moderate | 8
  Poor | 4

5. Secondary Outcome: Percentage of Patients Who Discontinue Lumigan® 0.01% Prior to 14 Weeks of Treatment
Description: Patients who discontinued Lumigan® 0.01% prior to 14 weeks was assessed as Yes or No.
Time Frame: 14 Weeks
Population: All patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 419
Percentage of Patients | 7.9

6. Secondary Outcome: Percentage of Patients Who Continue Lumigan® 0.01% Treatment
Description: Patients who will continue Lumigan® 0.01% after 14 weeks of treatment was assessed as Yes or No.
Time Frame: Week 14
Population: All patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 419
Percentage of Patients | 86.2

7. Secondary Outcome: Physician Assessment of Patient Compliance Compared to Previous Therapy
Description: Physician assessment of patient compliance compared to previous therapy was assessed on a 3-point scale (better, equal, and worse). The numbers of patients in each category are presented.
Time Frame: Week 14
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 184
Patients
  Better | 94
  Equal | 88
  Worse | 1
  Not Applicable | 1

8. Primary Outcome: IOP at Week 14
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eyes at Week 14.
Time Frame: Week 14
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 390
Millimeters of Mercury
  Right Eye | 15.92 (2.71)
  Left Eye (n=389) | 16.05 (2.73)

ADVERSE EVENTS:
Description: All enrolled patients were used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Lumigan® 0.01%
Serious Adverse Events (participants affected / at risk) | 0/419
Other Adverse Events (participants affected / at risk) | 57/419
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumigan® 0.01% (N=419)
Conjunctival Hyperaemia (Eye disorders) | 36
Eye Irritation (Eye disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.